CLINICAL TRIAL: NCT02715843
Title: Extended Treatment Access Study of MT-3724 for Subjects With Relapsed Non-Hodgkin's B-Cell Lymphoma Who Have Completed Phase I/Ib Study MT-3724_NHL_001_US
Brief Title: Extended Treatment Access Study of MT-3724 for Subjects With Relapsed Non-Hodgkin's B-Cell Lymphoma
Status: No longer available | Type: Expanded Access
Sponsor: Molecular Templates, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MT-3724_NHL_001_EXT_US
Record Dates: First submitted 2016-02-23; First posted 2016-03-22 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Non-Hodgkin's B-cell Lymphoma
Keywords: CD20; immunotoxin; NHL; non-Hodgkin's lymphoma; lymphoma; cancer; antibodies; immunotherapy; safety; pharmacokinetics; MT-3724; relapsed; refractory
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma; Neoplasms; Recurrence

INTERVENTIONS:
Drug: MT-3724 — Intravenous dosing M-W-F X 2 weeks; MT-3724 infusion over 2 hours on each dosing day over 4 week initial cycle and then 3 week repeat cycles for up to 5 total cycles.

SUMMARY:
This is an active treatment, extended access study open solely to those subjects who have successfully completed the Core and Repeat Dosing portions of the MT-3724_NHL_001_US clinical study and who, in the investigator's judgment, (i) have not had progressive disease while on MT-3724 treatment (i.e.; have shown a complete or partial response or stable disease), (ii) have experienced no clinical or laboratory toxicities that would contraindicate further MT-3724 dosing and (iii) have no acceptable and better alternative treatment available to them.

DETAILED DESCRIPTION:
Each treatment cycle will consist of 6 doses of MT-3724 to be administered over 12 days followed by at least 9 days of observation but longer intervals between dosing cycles will be allowed at the investigator's discretion (e.g., 6 doses of MT-3724 over 12 days followed by 16 days observation). Subjects in this extension study may continue to receive up to 6 additional cycles in the absence of clear disease progression or toxicity. If a subject achieves complete remission, two additional cycles will be attempted, after which dosing may be suspended prior to completion of the maximum 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must be adequately informed of all study procedures and fully consent to participation as demonstrated by signing the Informed Consent Form (ICF).
* Eligible subjects must require treatment for their NHL and have:

  * tolerated MT-3724 throughout the MT-3724_NHL_001_US Phase I/Ib study (Core and Repeat Dosing),
  * successfully completed the Core and Repeat Dosing portions of MT-3724_NHL_001_US Phase I/Ib study as defined by that protocol,
  * received no other treatment for their NHL since enrollment in the MT-3724_NHL_001_US Phase I/Ib study,
  * maintained stable disease or better throughout that study and
  * been assessed by the investigator to have no other acceptable and better treatment options available to them. The investigator must document in the potential subject's medical record that there are no other approved treatment options available and/or appropriate for the potential subject or that the potential subject has declined any other approved treatment options that me be available to them.
* Potential subjects must continue to meet the diagnostic criteria for B-Cell NHL that allowed them to be eligible for the MT-3724_NHL_001_US Phase I/Ib study.
* Potential subjects must have received all approved therapies known to provide clinical benefit for their disease subtype and for which they are eligible or must have refused these treatment options prior to consideration for continued compassionate use treatment with MT-3724 through enrollment in this protocol. In the case of subjects who have lymphomas for which high-dose chemotherapy and autologous stem cell transplantation (HD-ASCT) is considered a standard curative therapy, eligibility for MT-3724 compassionate use requires that the subject's disease relapsed after HD-ASCT, that the subject is not eligible for HD ASCT, or that the subject has refused HD-ASCT.
* Potential subjects with known central nervous system (CNS) metastases may be enrolled if they:

  * have previously been treated with radiotherapy for their CNS disease,
  * do not require chronic steroid therapy,
  * have had computed tomography or magnetic resonance imaging of the brain within 1 month of this study's entry that showed stable disease and
  * have no neurological symptoms (excluding Grade 1 or 2 neuropathy).
* Eastern Cooperative Oncology Group (ECOG) performance status of < 3
* Potential subjects should have measurable disease (any tumor mass of at least 1.5 cm) which has been documented to not have progressed during the MT-3724_NHL_001_US Phase I/Ib study and which can be followed during extended treatment for possible new disease progression.
* Potential subjects must be at least 9 days past their last course of MT-3724 treatment and have recovered from any side effects attributed to MT-3724 to at least Common Terminology Criteria for Adverse Events (CTCAE, v. 4.03; Appendix 4) Grade 2 prior to initiating additional cycles of MT-3724 through this compassionate use protocol. Subjects with pre-existing AEs at screening that are severe or life threatening by CTCAE grading should not be enrolled.
* Laboratory requirements:

  * Absolute neutrophil count (ANC) > 1,000 per microliter (μL)
  * Platelet count > 25,000/μL (The potential subject must be asymptomatic and the thrombocytopenia must be secondary to bone marrow infiltration by tumor and not secondary to increased platelet consumption or the effect of previous marrow suppressing treatment or infection.)
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin < 1.5 times upper limit of normal (ULN) (unless due to Gilbert's Disease)
  * Aspartate aminotransferase (AST; SGOT) and alanine aminotransferase (ALT; SGPT) < 2.5 times ULN or < 5x ULN if liver metastases are present
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 ml/min (either measured or estimated by the Cockcroft-Gault formula).
* Females of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to initiating dosing. Male and female subjects with reproductive potential must agree to use appropriate contraceptive methods while on study therapy and for 84 days following their last dose of study medication.

Exclusion Criteria:

* Patients who cannot comply with protocol requirements including clinic visits for intravenous infusions and birth control measures may not be enrolled.
* Female patients who are pregnant or are breast feeding.
* Potential patients with a history of another cancer other than basal cell carcinoma or cervical intraepithelial neoplasia (cervical cancer in situ) may not be enrolled unless it is documented that their previous cancer was treated, they have been disease free for five or more years prior to starting this study and they are in their doctor's judgment at less than 30% risk of relapse of this previous malignancy.
* Patients with a peripheral blood total lymphocyte count of higher than 25,000/mm3 may not be enrolled.
* Patients cannot have experienced a significant (CTCAE Grade 3 or 4 with or without neutropenia) infection within 2 weeks of their first dose of MT-3724.
* Patients are not eligible if they are using any other approved or investigational anti-neoplastic therapies or any other investigational therapies for any other reason.
* Patients may not be receiving systemic corticosteroid therapy at a prednisone dose > 20 mg/day (or steroid equivalent) within 2 weeks of starting study.
* Patients with uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months prior to start of study treatment, New York Heart Association (NYHA) Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, or cardiac amyloidosis may not be enrolled.
* Patients with a known history of drug abuse or any chronic neurologic, psychiatric, endocrine, metabolic, immunologic, hepatic or renal disease (including a history of hemolytic uremic syndrome) that in the opinion of the Investigator would adversely affect study participation.
* Patients with known active Hepatitis C, HIV or a present history of Hepatitis B
* Patients must not have received any vaccines for 28 days prior to administration of their first dose of MT-3724 and should not receive any vaccine during the study or within 28 days after their last dose of MT-3724.
* Patients with a suspected allergy or sensitivity to any component of MT-3724 drug preparation based upon known allergies to compounds of a similar class who have had an anaphylactic or other severe infusion reaction to human immunoglobulin or monoclonal antibody administration are n ot eligible.
* Patients who have had an allogeneic hematopoietic stem cell transplantation are not eligible.
* Patients who have had major surgery within 6 weeks prior to the first dose of study drug or have major surgery planned during the first 12 weeks after MT-3724 has finished.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas